CLINICAL TRIAL: NCT01364779
Title: Prevalence of Aspirin Resistance in Chronic Kidney Disease Patients
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Suzanne El-Sayegh, Nephrology Attending, Assoc. Chair of Medicine, Northwell Health
Other Study IDs: 10-025
Record Dates: First submitted 2011-05-27; First posted 2011-06-02 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Kidney Disease
Keywords: aspirin; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood draw
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective of the study is to determine the prevalence of aspirin resistance in chronic kidney disease patients. The secondary objectives are to determine possible risk factors contributing to aspirin resistance in this population.

DETAILED DESCRIPTION:
A cross-sectional of "aspirin resistance in hemodialysis patients" previously done in our institution showed that 23/66 (34.7%) hemodialysis patients were aspirin resistant. In a recent systematic review, renal impairment was associated with aspirin resistance . This association was seen in only two out of the twenty studies used in this meta-analysis . Both these studies are from the same center with a predominant Asian population. In this study we will try to evaluate the prevalence of aspirin resistance in CKD patient without being limited to a specific ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known structural kidney disease as evident by history or by urinalysis and CKD stage III or IV determined by MDRD formula and who are taking aspirin.

Exclusion Criteria:

* Younger than 18 years of age.
* Bleeding disorder or myeloproliferative disorders.
* Thrombocytopenia with platelets < 100.000.
* Malignancy.
* Acute hemorrhagic disease.
* A recent history of receipt of platelet glycoprotein IIb/IIIa blockers.
* Liver disease as evident by abnormal liver function and total bilirubin > 2mg/dl.
* use of anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the nephrology clinic at SIUH and the nephrology clinic at Staten Island rehab and the admitted patients who give consent.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
prevalence of aspirin resistance in chronic kidney disease patients | 2 years
  Blood drawn for the Accumetric test

SECONDARY OUTCOMES:
risk factors contributing to aspirin resistance in this population. | 2 years
  risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne El_Sayegh, MD, Principal Investigator — Staten Island University Hospital
Locations (1):
- staten island University Hospital nephrology clinic, Staten Island, New York, United States